CLINICAL TRIAL: NCT06614426
Title: The Efficacy of Electrolysis Decontamination with or Without Leukocyteplatelet Rich Fibrin (L-PRF) in the Surgical Treatment of Peri-implantitis Defects: a Randomized Controlled Trial
Brief Title: Surgical Treatment of Peri-implantitis Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer Hakam (Other)
Responsible Party: Sponsor-Investigator, Abeer Hakam, Assistant professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Organization: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBRU IRB-2024-563
Record Dates: First submitted 2024-09-18; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Peri Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (C): Conventional open flap debridement (Active Comparator): Conventional open flap debridement
  Interventions: Procedure: Control group (C)
- Test group 1 (T1): Open flap debridement using electrolysis decontamination (Experimental): Open flap debridement using (GalvoSurge® - Straumann)
  Interventions: Procedure: Test group 1 (T1)
- Test group 2 (T2): Open flap debridement using electrolysis decontamination combined with L-PRF (Experimental): Open flap debridement using (GalvoSurge® - Straumann) combined with L-PRF application
  Interventions: Procedure: Test group 2 (T2)

INTERVENTIONS:
Procedure: Test group 1 (T1) — Test group 1 (T1): Open flap debridement using electrolysis decontamination
  Arms: Test group 1 (T1): Open flap debridement using electrolysis decontamination
Procedure: Test group 2 (T2) — Test group 2 (T2): Open flap debridement using electrolysis decontamination combined with L-PRF application
  Arms: Test group 2 (T2): Open flap debridement using electrolysis decontamination combined with L-PRF
Procedure: Control group (C) — Conventional open flap debridement
  Arms: Control group (C): Conventional open flap debridement

SUMMARY:
The aim of this study is to evaluate the efficacy of implant surface decontamination using electrolysis cleaning system. And to evaluate the adjunctive use of L-PRF in promoting soft tissue healing and long-term stability of the peri-implant marginal bone in the surgical treatment of peri-implantitis.

DETAILED DESCRIPTION:
Research design

* Prospective, in which participants will be recruited and then followed up throughout a specified period of time.
* Randomized, parallel designed, concurrent controlled trial with participants randomly allocated to either control or test groups.
* Single-blinded as the outcome accessors will be blinded to the intervention.

Materials and Methods:

Patients attending Dubai Dental Hospital and requiring treatment of peri-implantitis will be invited to take part in this randomized controlled trial based on the following inclusion and exclusion criteria:

Inclusion criteria:

* Aged 18 or over.
* Require treatment of peri-implantitis (defined as the presence of bleeding and/or suppuration on gentle probing, probing depths of ≥ 6 mm, presence of bone loss beyond crestal bone level changes resulting from initial bone remodeling).
* Screw retained implant crown.
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion criteria

* History of surgical therapy of peri-implantitis.
* Peri-implant defects indicated for regenerative procedure (i.e. contained bony defect).
* Cement retained implant crown.
* Systemic/local antibiotics during the previous 6 months.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Smokers

The study will be conducted following the ethical standards of the Declaration of Helsinki in 1975, as revised in 2013 and the CONSORT statement will be used as a guideline in reporting this study.

Randomization, allocation concealment and blinding:

The participants will be randomly allocated to three equally sized groups using computer-generated numbers:

Control group (C): Conventional open flap debridement Test group 1 (T1): Open flap debridement using (GalvoSurge® - Straumann) Test group 2 (T2): Open flap debridement using (GalvoSurge® - Straumann) combined with L-PRF application

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Require treatment of peri-implantitis (defined as the presence of bleeding and/or suppuration on gentle probing, probing depths of ≥ 6 mm, presence of bone loss beyond crestal bone level changes resulting from initial bone remodeling).
* Screw retained implant crown.
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* History of surgical therapy of peri-implantitis.
* Peri-implant defects indicated for regenerative procedure (i.e. contained bony defect).
* Cement retained implant crown.
* Systemic/local antibiotics during the previous 6 months.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline (prior to surgical intervention), 3, 6, 12 and 24 months
  - Probing pocket depth: measured at baseline (prior to surgical intervention), 3, 6, 12 and 24 months using a manual periodontal probe.

SECONDARY OUTCOMES:
Presence or absence of plaque, bleeding on probing and suppuration | Baseline (prior to surgical intervention), 3, 6, 12 and 24 months
  Presence or absence of plaque, bleeding on probing and suppuration: measured at baseline (prior to surgical intervention), 3, 6, 12 and 24 months using a manual periodontal probe
Peri-implant marginal bone level | Baseline (prior to surgical intervention), 12 and 24 months
  - Peri-implant marginal bone level: measured at baseline (prior to surgical intervention), 12 and 24 months using standardized peri-apical radiographs.
Peri-implant soft tissue level | Baseline (prior to surgical intervention), 3, 6, 12 and 24 months
  - Peri-implant soft tissue level: measured at baseline (prior to surgical intervention), 3, 6, 12 and 24 months using a manual periodontal probe.
Peri-implant soft tissue thickness (Phenotype) | Baseline (prior to surgical intervention), 3, 6, 12 and 24 months
  - Peri-implant soft tissue thickness (Phenotype): measured at baseline (prior to surgical intervention), 3, 6, 12 and 24 months using an endodontic spreader at 3 points.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamzacebi B, Oduncuoglu B, Alaaddinoglu EE. Treatment of Peri-implant Bone Defects with Platelet-Rich Fibrin. Int J Periodontics Restorative Dent. 2015 May-Jun;35(3):415-22. doi: 10.11607/prd.1861. PMID 25909530